CLINICAL TRIAL: NCT05610904
Title: Evaluation of a Machine Learning Based Anastomotic Leakage Prediction Model After Anterior Resection for Rectal cancer-a Multicenter, Prospective, Randomized Controlled Study
Brief Title: Evaluation of AL Prediction for Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhang, professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHALP001
Record Dates: First submitted 2022-10-30; First posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Anastomotic Leak Rectum
Keywords: Anastomotic Leak; rectal cancer; machine learning
MeSH Terms: conditions — Anastomotic Leak; Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgeon evaluation (No Intervention)
- Surgeon combining with model evaluation (Experimental)
  Interventions: Diagnostic Test: Prediction model evaluation

INTERVENTIONS:
Diagnostic Test: Prediction model evaluation — a machine learning based anastomotic leakage prediction model
  Arms: Surgeon combining with model evaluation

SUMMARY:
Anastomotic leakage is one of the most serious postoperative complications of low rectal cancer, with an incidence of 3%-21%. The occurrence of anastomotic leakage is related to many factors, and the occurrence of anastomotic leakage can be predicted by building a prediction model. Most of the anastomotic leakage prediction models constructed in the past are nomograms, which have limitations in the fitting of model creation. In the previous study, the center took the lead in building a random forest anastomotic leakage prediction model based on machine learning. This study intends to prospectively enroll patients with rectal cancer undergoing anterior abdominal resection and use their clinical data to prospectively verify the efficacy of the anastomotic leakage prediction model, and further improve and promote the prediction model.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-75 years
2. Adenocarcinoma confirmed by pathology
3. Colonoscopy or imaging examination confirmed that the distance between the lower edge of the tumor and the anal edge was less than or equal to 12cm
4. Preoperative imaging diagnosis was cTxNxM0
5. No local complications (no obstruction, incomplete obstruction, no massive active bleeding, no perforation, abscess formation, and no invasion of adjacent organs)
6. The hematopoietic functions of heart, lung, liver, kidney and bone marrow meet the requirements of surgery and anesthesia
7. Voluntarily sign the informed consent form

Exclusion Criteria:

1. Previous history of malignant tumor
2. Simultaneous multiple primary colorectal cancer
3. Previous multiple abdominal and pelvic surgeries or extensive abdominal adhesions
4. Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc., requiring emergency surgery
5. Patients with familial adenomatous polyposis and active inflammatory bowel disease
6. A history of severe mental illness
7. pregnant or lactating women
8. Patients with uncontrolled infection before operation
9. The investigator did not consider the patient to be eligible for the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2022-12-10 (Estimated); Primary Completion 2024-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Accuracy of stoma implementation | 1 months after surgery
  Accuracy of stoma implementation: the number of anastomotic leakage patients with stoma and none anastomotic leakage patients without stoma to the number of total patients.

SECONDARY OUTCOMES:
Sensitivity and specificity in the prediction of anastomotic leakage | 1 months after surgery
Grade C leakage rate | 1 months after surgery
Preventive stoma rate | 1 months after surgery
Rate of stoma reverse | 3-6 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Colorectal Surgery in Changhai Hospital, Shanghai, Shanghai Municipality, China